CLINICAL TRIAL: NCT06954727
Title: China Pulmonary Vascular Disease Intervention Diagnosis and Management Study-A Quality Control on Right Heart Catheterization
Brief Title: China Pulmonary Vascular Disease Intervention Diagnosis and Management Study-right Heart Catheterization
Acronym: CHA-RHC
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Professor, China-Japan Friendship Hospital
Other Study IDs: CHALLENGE-RHC; 2023YFC2507200 (Other Grant/Funding Number: The National Key Research and Development Program of China)
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Hypertension; Pulmonary Embolism (Diagnosis); Pulmonary Arterial Hypertension; Right Heart Catheterization
Keywords: right heart catheterization; pulmonary hypertension; pulmonary arterial hypertension; pulmonary vascular disease
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Embolism; Disease; Pulmonary Arterial Hypertension | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who underwent right heart catheterization: The study population consists of patients who underwent right heart catheterization for the first time due to dyspnea or suspected pulmonary hypertension. No intervention.
  Interventions: Other: No intervention; Observational study

INTERVENTIONS:
Other: No intervention; Observational study — No intervention; observational study

SUMMARY:
Right heart catheterization(RHC) plays a crucial role in the diagnosis and treatment of pulmonary vascular diseases(PVD). In China, the lack of equipment and technical expertise has historically limited the implementation of RHC, thereby greatly restricting the diagnosis and treatment of RVD. In recent years, with improvements in these issues, more hospitals have acquired the capability to perform RHC. The purpose of this study is to conduct quality control of RHC across multiple pulmonary hypertension(PH) centers in China. The study population consists of patients who underwent RHC for the first time due to dyspnea or suspected PH. This study retrospectively and prospectively collects multicenter RHC data, with the main quality control contents including indications for the procedure, collection and analysis of hemodynamic data, diagnosis and treatment, and long-term management of patients.

DETAILED DESCRIPTION:
This study is led by the China-Japan Friendship Hospital and will be conducted across approximately 30 pulmonary hypertension centers in China. It is an observational cohort study without interventional treatment. Eligible participants are patients aged 14 years or older who undergo right heart catheterization due to dyspnea or suspected pulmonary hypertension. After study initiation, investigators at each center will enroll eligible patients and collect baseline data, hemodynamic parameters from right heart catheterization, diagnostic classification of pulmonary hypertension, and treatment plans. Patients will receive routine follow-up at their respective centers, and investigators will gather follow-up data according to the study protocol. All de-identified data will be recorded in an Electronic Data Capture (EDC) system. A dedicated data management team will oversee data management, quality control, and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent right heart catheterization for the first time due to dyspnea or suspected pulmonary hypertension
* Age ≥14 years old

Exclusion Criteria:

* Vital data missing
* Did not sign informed consent or did not agree to follow-up

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent right heart catheterization for the first time due to dyspnea or suspected pulmonary hypertension and age over 14 years old
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
3-month all cause death | 3 month
  3-month all cause death

SECONDARY OUTCOMES:
dignosis and type of pulmonary hypertension | 1 month
  dignosis and type of pulmonary hypertension according to latest guidelines
1-year all cause death | 1 year
  1-year all cause death

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Zhai, PhD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
We retain the property rights to the patient-level data, and therefore will not share this data. We plan to publish the study results and provide aggregate data when necessary.